CLINICAL TRIAL: NCT00252187
Title: Cardiac Hormone Replacement With BNP in Heart Failure: A Novel Therapeutic Strategy
Brief Title: Cardiac Hormone Replacement With Brain Natriuretic Peptide (BNP) in Heart Failure
Acronym: SubqBNP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Horng Chen (Other)
Collaborators: American Heart Association (Other); Scios, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Horng Chen, MD, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69-00; R01HL036634 (NIH); R01HL084155 (NIH); P01HL076611 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Congestive Heart Failure; Cardiomyopathy
Keywords: Heart failure; Natriuretic peptides; B-type natriuretic peptide; Kidney; Nesiritide; Natrecor; CHF
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-type Natriuretic Peptide (BNP) (Active Comparator): BNP (nesiritide) administered subcutaneously twice daily for 8 weeks at 10 mcg/kg.
  Interventions: Drug: B-type Natriuretic Peptide (BNP)
- Placebo (Placebo Comparator): Placebo self-administered subcutaneously twice daily for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: B-type Natriuretic Peptide (BNP) — BNP hormone self-administered subcutaneously twice daily for 8 weeks at 10 mcg/kg.
  Other Names: Nesiritide
  Arms: B-type Natriuretic Peptide (BNP)
Other: Placebo — Placebo self-administered subcutaneously twice daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of subcutaneous injection of Human BNP (nesiritide), a hormone produced by the heart, on the pumping ability of the heart, kidney function, and hormonal function in persons with heart failure.

DETAILED DESCRIPTION:
The cardiac hormone brain natriuretic peptide (BNP) plays an important role in the pathophysiology of congestive heart failure (CHF). Studies have established that BNP mediates natriuresis, renin and aldosterone (RAAS) inhibition, vasodilation and lusitropism. Acute cardiac hormone replacement with intravenous infusion of BNP has been shown to possess potent vasodilating actions in humans with acute decompensated CHF resulting in improvement of clinical symptoms. Natrecor (nesiritide) a sterile, purified preparation of human BNP is approved by the FDA for intravenous administration in the treatment of patients with acute decompensated congestive heart failure. However, chronic cardiac hormone replacement with BNP as therapeutic strategy in CHF has been limited by the need to administer BNP intravenously. The objective of this study is to define the cardiorenal and humoral actions of short term (eight weeks) chronic cardiac hormone replacement with subcutaneous (SQ) BNP in human NYHA class II-III CHF. Systolic and diastolic function, left ventricular remodeling as assessed by its volume, renal function, neurohumoral profiling and exercise capacity will be assessed prior to and after eight weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Resting left ventricular ejection fraction (LVEF) of 35% or less (determined within 48 months of recruitment by echocardiography, multiple gate acquisition scan (MUGA) or left ventriculogram.)
3. New York Heart Association (NYHA) Class I (with previous symptoms of heart failure), Class II and III
4. Female subjects not menopausal or surgically sterilized will need to have a negative pregnancy test the day before the study day and be on contraception.

Exclusion Criteria:

1. Myocardial infarction (MI) within 3 months of screening.
2. Unstable angina within 14 days of screening, or any evidence of myocardial ischemia.
3. Valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis.
4. Sustained ventricular tachycardia (VT) or ventricular fibrillation (V-fib) within 14 days of screening.
5. Second or third degree atrioventricular (AV) block without a permanent cardiac pacemaker.
6. Cerebrovascular accident (CVA) within 3 months of screening, or other evidence of significantly compromised central nervous system (CNS) perfusion.
7. Serum creatinine of >3.0 mg/dL.
8. Serum sodium of <125 milliequivalents per decaLiter (mEq/dL) or > 160 mEq/dL.
9. Serum potassium of < 3.5 mEq/dL or > 5.2 mEq/dL.
10. Serum digoxin level of > 2.0 ng/ml.
11. Systolic pressure of <85 mmHg immediately prior to the first injection of study drug/placebo.
12. LVEF > 35% by within 24 months of screening.
13. Unable to self-administer subcutaneous injection twice a day.
14. Diagnosed with AIDS or known positive HIV titer.
15. Other acute or chronic medical conditions or laboratory abnormality, which may increase the risks, associated with study participation or may interfere with interpretation of the data.
16. Received an investigational drug within 1 month prior to dosing.
17. Unable to undergo cardiac magnetic resonance imaging (MRI). Contraindications to MRI include pacemaker or defibrillator, pregnant women, atrial fibrillation or other arrhythmia, cerebral aneurysm clips, or severe claustrophobia.
18. In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reasons.
19. Patient in atrial fibrillation or who have a pacemaker or implantable cardioverter defibrillator (ICD)
20. Hemoglobin < 10g/dl.
21. Patients with an allergy to iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2000-01; Primary Completion 2008-07 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Chen HH, Glockner JF, Schirger JA, Cataliotti A, Redfield MM, Burnett JC Jr. Novel protein therapeutics for systolic heart failure: chronic subcutaneous B-type natriuretic peptide. J Am Coll Cardiol. 2012 Dec 4;60(22):2305-12. doi: 10.1016/j.jacc.2012.07.056. Epub 2012 Nov 1. PMID 23122795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2003 to May 2008 at the Mayo Clinic in Rochester, Minnesota.
Groups:
- B-type Natriuretic Peptide (BNP): BNP (nesiritide) hormone self-administered subcutaneously twice daily for 8 weeks at 10 mcg/kg.
Period: Overall Study
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Started | 24 | 21
Completed | 20 | 20
Not Completed | 4 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 13 | 10 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 65 (11) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 20 | 13 | 33
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45
Blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure (SBP) the top number and diastolic blood pressure (DBP)the bottom number in a blood pressure reading, are measured in millimeters of mercury (mmHg) on a scale.
  mmHg
    Systolic blood pressure | 131 (18) | 127 (17) | 129 (17)
    Diastolic blood pressure | 72 (11) | 72 (14) | 72 (12)
New York Heart Association (NYHA) CHF Classification [Number; unit: participants] — NYHA classifications of various stages of Congestive Heart Failure (CHF) help determine the severity. Class I-No symptoms at any level of exertion & no limitation in ordinary physical activity. Class II-Mild symptoms and slight limitation during regular activity. Comfortable at rest. Class III-Noticeable limitation due to symptoms, even during minimal activity; Comfortable only at rest. Class IV-Severe limitations. Symptoms even while at rest. Note: The sum of categorized subjects will not equal the total number of participants enrolled in each arm, because only Class II & III were reported.
  participants
    NYHA CHF Class II | 13 | 10 | 23
    NYHA CHF Class III | 2 | 1 | 3
Left Ventricle Ejection Fraction (Echo) [Mean (Standard Deviation); unit: Percentage] — Left Ventricle Ejection Fraction (LVEF)is a clinical parameter used by cardiologists to describe how well the heart is pumping. LVEF is a measure of the amount of blood pumped out of the lower chamber (ventricle) of the heart during a heartbeat, measured by echocardiography. A normal LVEF ranges from 55-70%. A LVEF of 65, for example, means that 65% of the total amount of blood in the left ventricle is pumped out with each heartbeat.
  Percentage | 32 (9) | 31 (7) | 31 (8)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Heart rate (HR) is a measure of how many times the heart beats per minute.
  beats per minute | 65 (13) | 68 (12) | 67 (13)
Plasma BNP [Median (Inter-Quartile Range); unit: picograms/milliliter] — B-type natriuretic peptide (BNP) is a cardiac hormone that affects cardiovascular function.
  picograms/milliliter | 51 [18 to 102] | 63 [10 to 318] | 53 [12 to 153]
Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — Glomerular Filtration Rate (GFR) is a measure of the flow rate or speed the kidney filters fluid, measured in milliliters per minute per 1.73 m^2 of body-surface area. A lower GFR means the kidney is not filtering normally. An estimated GFR of less than 60 ml/min/1.73 m^2 of body-surface area is considered to be impaired kidney function.
  ml/min/1.73 m^2 | 73 (22) | 77 (21) | 75 (22)
History or concomitant medical conditions [Number; unit: participants] — Because participants may have none, one, or more than one medical history or concomitant medical condition, the sum of the history categories will not be the same as the overall number of participants in a given arm of the study.
  participants
    History of peripheral vascular diseases | 2 | 1 | 3
    History of chronic obstructive pulmonary disease | 3 | 1 | 4
    History of Coronary Artery Disease | 11 | 11 | 22
    History of hypertension | 10 | 17 | 27
    History of arrythmia | 5 | 4 | 9
    History of smoking | 10 | 8 | 18
    History of diabetes | 11 | 7 | 18
    History of high cholesterol | 15 | 17 | 32
Concomitant Medication(s) [Number; unit: participants] — The sum of subjects taking a given class of medication will not equal the overall number of participants per arm, because all subjects would possibly not be taking all medication classes.
  participants
    ACE I inhib, Angio II receptor blocker or nitrates | 23 | 20 | 43
    Digoxin | 8 | 9 | 17
    Beta blocker | 23 | 20 | 43
    Coumadin | 3 | 1 | 4
    Antiarrhythmics | 5 | 0 | 5
    Diuretic (loop) | 18 | 15 | 33
    Diuretic (thiazide) | 4 | 3 | 7
    Diuretic (potassium sparing) | 5 | 4 | 9
    Diuretic (Thiazide) | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular (LV) Volume Index at 8 Weeks
Description: LV volume was measured for systolic volume and diastolic volume using a cardiac Magnetic Resonance Imaging (MRI) scan. All cardiac MRI images were reviewed by an independent cardiologist in a blinded fashion.
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
ml/m^2
  End-systolic LV volume index | -5.2 (13) | 5.8 (9.6)
  End-diastolic LV volume index | -10.0 (15.4) | 6.1 (12.4)
Statistical Analysis 1: Comparison: B-type Natriuretic Peptide (BNP) vs Placebo; Change in end systolic LV volume index compared between two groups; Test type: Superiority or Other; p = 0.004, Chi-squared
Statistical Analysis 2: Comparison: B-type Natriuretic Peptide (BNP) vs Placebo; Change in LV end diastolic volume was compared between two groups; Test type: Superiority or Other; p = 0.001, Chi-squared

2. Secondary Outcome: Change in Left Ventricular (LV) Filling Pressure at 8 Weeks
Description: Filling pressure determined by ratio of E/e' [Echocardiograph Doppler mitral inflow velocity (E) to mitral annulus tissue Doppler velocity (e') ratio]
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: E/e'
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
E/e' | -2.3 (2.5) | 1.1 (3.1)
Statistical Analysis 1: Comparison: B-type Natriuretic Peptide (BNP) vs Placebo; Test type: Superiority or Other; p = 0.001, Chi-squared

3. Secondary Outcome: Change in Plasma Renin Activity at 8 Weeks
Description: Plasma renin is synthesized within circulation or at tissue sites, causing vasoconstriction or vasodilation.
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter per hour
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
nanograms per milliliter per hour | -3.5 (7.1) | 2.3 (4.8)

4. Secondary Outcome: Change in Renal Function as Measured by Glomerular Filtration Rate (GFR) at 8 Weeks
Description: Kidney function was measured by GFR determined by iothalamate clearance. Glomerular filtration rate describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body-surface area. A lower GFR means the kidney is not filtering normally.
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2 of body-surface area
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
ml/min/1.73 m^2 of body-surface area | 6.9 (14.2) | -2.8 (24.8)
Statistical Analysis 1: Comparison: B-type Natriuretic Peptide (BNP) vs Placebo; Test type: Superiority or Other; p = 0.14, Chi-squared

5. Primary Outcome: Change in Left Ventricular (LV) Mass Index at 8 Weeks
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mg/m^2
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
mg/m^2 | -4.4 (9.8) | 6.2 (12.9)
Statistical Analysis 1: Comparison: B-type Natriuretic Peptide (BNP) vs Placebo; Test type: Superiority or Other; p = 0.006, Chi-squared

6. Secondary Outcome: Change in Heart Rate at 8 Weeks
Description: Heart rate was measured when MRI was performed
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
beats per minute | -1.6 (8.3) | -0.9 (7.2)

7. Secondary Outcome: Change in Blood Pressure at 8 Weeks
Description: Blood pressure was measured during the MRI
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
mmHg
  Change in systolic blood pressure | -4.9 (22.2) | 4.5 (17.7)
  Change in diastolic blood pressure | -2.4 (8.5) | 0.9 (12.1)

8. Secondary Outcome: Change in Left Ventricular Ejection Fraction at 8 Weeks
Description: Left Ventricle Ejection Fraction (LVEF)is a clinical parameter used by cardiologists to describe how well the heart is pumping. LVEF is a measure of the amount of blood pumped out of the lower chamber (ventricle) of the heart during a heartbeat, measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline and 8 weeks
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | B-type Natriuretic Peptide (BNP) | Placebo
Number analyzed (Participants) | 20 | 20
percentage | 0.0 (7.5) | -1.1 (4.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 8 week study period
Groups:
- BPN Group: BNP (nesiritide) administered subcutaneously twice daily for 8 weeks at 10 mcg/kg.
Arm/Group | BPN Group | Placebo
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/21
Other Adverse Events (participants affected / at risk) | 20/24 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPN Group (N=24) | Placebo (N=21)
hypotension (Cardiac disorders) | 1 (1) | 0 (0) — 3 subjects in the BNP group developed hypotension (defined by systolic BP <85 mmHg)or had symptoms of light-headedness or visual disturbances during the baseline visit in the Clinical Research Unit. All recovered w/ adjusted position & fluids.
lightheadedness (Cardiac disorders) | 1 (2) | 0 (0)
visual disturbances (Eye disorders) | 1 (1) | 0 (0)
worsening heart failure symptoms (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | BPN Group (N=24) | Placebo (N=21)
Lightheadedness (Cardiac disorders) | 3/20 (3) | 0/20 (0)
Shortness of Breath and Fatigue (Cardiac disorders) | 3/20 (3) | 7/20 (7)
Injection site sting/itchy (Skin and subcutaneous tissue disorders) | 4/20 (4) | 3/20 (3)
Flu-like symptoms (General disorders) | 1/20 (1) | 2/20 (2)
Flushing (Blood and lymphatic system disorders) | 3/20 (3) | 1/20 (1)
Loose stools (Gastrointestinal disorders) | 2/20 (2) | 0/20 (0)
Atrial Fibrillation (Cardiac disorders) | 0/20 (0) | 1/20 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1/20 (1) | 1/20 (1)
Edema (Blood and lymphatic system disorders) | 1/20 (1) | 0/20 (0)
GI bleed prior to study drug administration (Gastrointestinal disorders) | 1/20 (1) | 0/20 (0)
Increased voiding (Renal and urinary disorders) | 1/20 (1) | 0/20 (0)
Choledocholithiasis (Hepatobiliary disorders) | 0/20 (0) | 1/20 (1) — Gall stone in bile duct was accompanied by fever and elevated liver function test result.
Head congestion and productive cough (Infections and infestations) | 0/20 (0) | 1/20 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No